CLINICAL TRIAL: NCT03244722
Title: Maternal Metabolic and Molecular Changes Induced by Preconception Weight Loss and Their Effects on Birth Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Amy E Rothberg, Project Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00124673; 1R01DK124862 (NIH)
Record Dates: First submitted 2017-08-05; First posted 2017-08-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Familial; Pregnancy Related
MeSH Terms: conditions — Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Obese - Very low energy diet (VLED) (Other): Participants will adopt a very-low energy diet
  Interventions: Dietary Supplement: Very-low energy Diet (VLED)
- Obese - Standard of care (SOC) (Other): Participants will receive the standard of care for obese women looking to become pregnant.
  Interventions: Other: Standard of care (SOC)
- Lean - Standard of care (SOC) (Other): Participants will receive the standard of care for lean women looking to become pregnant.
  Interventions: Other: Standard of care (SOC)

INTERVENTIONS:
Dietary Supplement: Very-low energy Diet (VLED) — Structured, intensive dietary intervention using liquid meal replacements aimed at providing 800 kcal/day with a weight loss goal of 15% from baseline
  Arms: Obese - Very low energy diet (VLED)
Other: Standard of care (SOC) — Standard consultation with registered dietitian to determine appropriate caloric deficit for a low calorie diet, education and advice to achieve weight loss in obese women. Standard of care for normal weight women
  Arms: Lean - Standard of care (SOC); Obese - Standard of care (SOC)

SUMMARY:
Our hypothesis is that aggressive preconception weight loss in obese women will improve the metabolic health of the mother and the intrauterine environment. An optimized developmental environment will normalize fetal growth and improve clinical fetal and infant outcomes, and theoretically reduce future susceptibility to obesity and cardiometabolic disease.

DETAILED DESCRIPTION:
Further, our hypothesis is that the metabolic profiles in the mother and infant cord blood and epigenetic profiles in cord blood leukocytes will be improved in the very-low energy diet (VLED) group compared to standard practice nutrition counseling and support (SOC) group and approach the profiles found in normal weight (LEAN) individuals. We will relate these changes to the changes in the offspring clinical profiles. With these data in hand, we will develop a model to understand the potential molecular markers associated with offspring size and adiposity at birth, risk factors for later onset non-communicable diseases. We will use these insights to define, adopt and implement future interventions that mitigate the downstream risk of adiposity and cardiometabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 ≤ 45 for obese participants OR
* BMI ≤ 25 for healthy body weight participants
* No known infertility
* No known risk factors for tubal disease

Exclusion Criteria:

* Significant medical co-morbidities (e.g. heart, kidney, liver, autoimmune disease)
* Significant anemia
* Cancer other than minor skin cancers
* Conditions that would complicate pregnancy
* Recent use of anti-obesity drugs or appetite suppressants
* Previous bariatric surgery
* Endometriosis AFS (American Fertility Society classification class III or IV)
* Progesterone > 10 IU/ml
* Current pregnancy
* Use of sperm donor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Preconception weight loss | Baseline to post dietary intervention (16 weeks)
  Primary pre-specified outcome is BMI change (kg/m2) after dietary intervention. Trained staff will measure height and weight to the nearest .1cm and .1kg using a wall-mounted, precision stadiometer and calibrated digital scale. BMI will be calculated (kg/m2).
Metabolome and inflammatory markers | Delivery
  Multivariate computational models will assess the association of maternal and neonate metabolite and inflammatory markers to fetal growth and newborn weight (g) and adiposity (g).
Offspring body fat mass | Delivery
  Percentage body fat (adiposity) in the offspring of women randomized to Very Low Energy Diet (VLED) compared to those randomized to Standard of Care (SOC). Body composition will be assessed by PeaPod (fat mass in grams).
Cord blood related to neonate outcomes | Before and after dietary intervention (16 weeks), delivery
  The maternal metabolome (~metabolites) will be related to neonate adiposity, gestational weight gain, pregnancy complications, and intrauterine fetal growth rate.
DNA methylation | Delivery
  Differences in site-specific DNA methylation (~450,000 sites) in offspring cord blood mononuclear cells between the Standard of Care (SOC), Very Low Energy Diet (VLED) and lean groups will be assessed.

SECONDARY OUTCOMES:
Participant waist circumference in centimeters | Baseline and post dietary intervention (16 weeks), each trimester of pregnancy (between 8-12 weeks, between 18-22 weeks, and between 28-34 weeks)
  The change in waist circumference (cm) will be assessed using a retractable, soft nylon measuring tape.
Fetal growth will be assessed by ultrasound | Each trimester of pregnancy (between 8-12 weeks, between 18-22 weeks, and between 28-34 weeks)
  Gestational sac dimensions (mm), fundal height (mm), biparietal diameter (mm), head circumference (mm), and waist circumference (mm) will be assessed through ultrasound to determine fetal growth.
Infant length and weight | Delivery to 12 month follow-up
  Trained staff will measure infant length and weight to the nearest .1cm and .1kg using an infant length board and digital infant scale at delivery, 2-, 4-, 6-, 9-, and 12-months. Ponderal index will be calculated and used to assess change in growth.
Metabolite levels | Each trimester of pregnancy (between 8-12 weeks, between 18-22 weeks, and between 28-34 weeks), delivery
  Relationships between metabolite levels (~2000 metabolites) in maternal blood at each trimester and cord blood mononuclear cell DNA methylation will be compared

OTHER OUTCOMES:
Mode of delivery | Delivery
  Categorical as caesarean or vaginal delivery
Fetal growth abnormalities | Each trimester of pregnancy (between 8-12 weeks, between 18-22 weeks, and between 28-34 weeks)
  Categorical as miscarriage, intrauterine growth restriction (IUGR), fetal demise, fetal anomalies
Maternal diagnosis | Each trimester of pregnancy (between 8-12 weeks, between 18-22 weeks, and between 28-34 weeks), delivery
  Categorical as maternal cardiac dysfunction, maternal proteinuria, maternal sleep apnea, fatty liver disease, gestational diabetes, preeclampsia, indicated preterm birth date, failed trial of labor, endometritis, venous thrombosis, COVD-19, surgical wound complications, postpartum anemia, postpartum depression, early termination of breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Rothberg, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No